CLINICAL TRIAL: NCT05821881
Title: Effects of Discontinuation of Levothyroxine Treatment in Older Adults: a Self-controlled Study
Brief Title: REduction of LEvothyroxine in Adults; a SElf Controlled Study
Acronym: RELEASE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, jgussekloo, Professor in primary care, Leiden University Medical Center
Other Study IDs: NL69753.058.19; NL7978 (Registry Identifier: Netherlands Trial Register); 839110026 (Other Grant/Funding Number: ZonMW HGOG)
Record Dates: First submitted 2023-04-05; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Hypothyroidism
Keywords: humans; aged; aged, 80 and over; thyroxine; deprescriptions; observational study; thyroid diseases; hypothyroidism; quality of life; health status; personal satisfaction; general practitioners
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Discontinuation of levothyroxine treatment — Step-wise reduction of levothyroxine treatment guided by thyroid function and symptoms

SUMMARY:
Many older persons use the thyroid hormone levothyroxine which is often continued for life. Scientifically, there is much uncertainty whether simple continuation is the optimal approach. The goal of this self-controlled observational study is to investigate how many participants of 60 years and older who are currently using levothyroxine, can be successfully withdrawn from levothyroxine treatment, either fully or partially, while maintaining a normal thyroid function (defined as a free T4 level within the reference range and a thyroid stimulating hormone [TSH] level <10 mU/L), 52 weeks after the start of the discontinuation.

Levothyroxine treatment is discontinued gradually guided by the participant's general practitioner, using a step-wise approach with regular monitoring of thyroid function. In addition, the effects of discontinuation of levothyroxine on thyroid-specific quality of life and general health will be studied using questionnaires.

DETAILED DESCRIPTION:
Study design - This is a self-controlled trial investigating the stepwise discontinuation of levothyroxine treatment in adults aged 60 years and older with a follow-up of 1 year. Outcomes will be measured 12 weeks before the start of discontinuation, at the start of discontinuation, at 6 weeks, at the end of discontinuation, and after 52 weeks. The outcomes will be compared within participants.

Study phases

* This study consists of 3 phases: a control phase of 12 weeks (T-12 to T0), the discontinuation phase (minimum of 6 weeks, maximum of 36 weeks; T0 to Tx), and a follow-up phase (from the end of discontinuation till 52 weeks after the start of discontinuation; Tx to T52).
* Control phase: participants enter the study during a control period with pre-baseline measurements of thyroid function and secondary outcome parameters to determine natural variation after which treatment with levothyroxine is continued per usual care for at least 12 weeks. Participants with a pre-baseline TSH level ≥10 mU/L do not proceed to the discontinuation phase.
* Discontinuation phase: this phase starts with baseline measurements of thyroid function and secondary outcome parameters, followed by a consultation of the participant with their GP during which discontinuation of levothyroxine is initiated, except when TSH level ≥10 mU/L. Levothyroxine is discontinued stepwise, and at intervals of ≥ 6 weeks to ascertain a steady-state concentration has been reached before the following control visit. During each '6-week' visit, the GP evaluates thyroid function and symptoms with the participant. Upon agreement, the daily dose of levothyroxine can then be lowered provided thyroid function is within the predefined limits, i.e. a normal fT4 and TSH < 10 mU/L. With each step, the dose of levothyroxine is reduced by approximately 25 mcg. The discontinuation phase ends after the evaluation of complete withdrawal of the levothyroxine treatment (i.e. 6 weeks after the final discontinuation step). Secondary outcome parameters are collected at the first '6-week' visit and the end of discontinuation.
* Follow-up phase: this phase ends with a final visit 52 weeks after the start of the discontinuation phase and includes the assessment of thyroid function, current dose of levothyroxine, and secondary outcome parameters.

Sample size

- The sample size calculation is based on the primary outcome, the proportion of participants successfully stopping levothyroxine treatment between baseline and final follow-up at 52 weeks. The investigators estimated a proportion of 50% of the participants would successfully discontinue levothyroxine treatment. A sample size of 385 participants was chosen because this allows to estimate the expected proportion of 50% with a 95% confidence interval of which the lower and upper limit is expected to deviate by 5 percentage points from the found percentage (i.e. 45% to 55% when the found percentage is indeed 50%). Taking a maximum of 25% loss to follow up into account over the duration of 15 months (exclusion at T-12 when TSH level ≥ 10 mU/L and/or fT4 below reference range, withdrawal, moving away, or death between T-12 and T52) a maximum of 513 participants will be recruited.

Data analysis

* GPs transfer participants' data after each visit using a validated electronic data capture (EDC) system (Castor EDC). Questionnaires are completed on paper or electronically (Castor EDC). All participant data are coded. Only the principal investigators and the research team have access to the key to these codes. The handling of personal data complies with the European General Data Protection Regulation. Database validation checks are run routinely and are tracked and escalated as appropriate.
* To determine the proportion of the population that can be withdrawn from levothyroxine treatment, categorical data involving measurements at baseline and final follow-up will be analyzed. Univariable and multivariable logistic regression analyses will be performed to assess factors that are associated with successful discontinuation of levothyroxine treatment. To estimate the effect of discontinuation on secondary outcome parameters measured at baseline and/or final follow-up, descriptive, univariable and multivariable analyses will be performed for the overall group and for the group of participants who successfully discontinued levothyroxine. Measurements pre and post discontinuation will be compared. Variations in thyroid function, thyroid-related quality of life, treatment satisfaction for levothyroxine, general health, and participant's attitude toward deprescribing will be determined using pre-baseline and baseline measurements. All analyses will be carried out with the population of participants who enrolled at baseline (T0). Participants that experience intercurrent events not related to the study procedure resulting in missing data at final follow-up will be excluded. Primary and secondary analyses will be repeated with all participants who enrolled at baseline who have data for the outcome variable of interest and have had their final follow-up visit. Statistical significance for the primary outcome requires P ≤ 0.05.

Safety and monitoring

* Withdrawal. Participants can withdraw their consent for involvement in the study at any time, without an obligation to justify the decision, and without consequences for their usual care. The research team can advise withdrawing participants from the intervention if it is deemed to be in the best interest of the participant. Participants who withdraw from the study are not replaced. The Data Safety and Monitoring Board (DSMB) can advise to stop the study.
* (Serious) adverse events. All adverse events reported spontaneously by the participant or their general practitioner (GP) are recorded and followed up. If complaints are reported during the discontinuation phase, these will be assessed by the research nurse. It is at the discretion of the GP to decide to either continue the withdrawal of levothyroxine or to maintain or increase the dosage. Serious adverse events are sought out actively and reported to the sponsor, the accredited Medical Ethics Committee (MEC), and competent authority using electronic case report forms.
* Monitoring. At regular intervals, the DSMB advises the study project group and sponsor (Leiden University Medical Center [LUMC]) whether it is safe and appropriate to continue the study. Periodic routine reports on the progress of the study are sent to the DSMB for review. Serious adverse events are reported immediately. No interim analyses for efficacy or futility will be performed. The DSMB meets at least 5 times and is composed of medical experts and a biostatistician without any involvement in the study as investigators or as study participant care physicians. Annual study monitoring visits are conducted by an independent clinical research associate (LUMC) according to a study-specific monitoring plan. A summary of the study progress is submitted to the MEC yearly, including the date of inclusion of the first participant, the number of participants included, the number of participants that have completed the trial, serious adverse events, and amendments.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 years or over (≥ 60 years)
2. Using any levothyroxine mono-therapy medicament (ATC: H03AA01) continuously for a minimum of 1 year with stable dose of levothyroxine.

Exclusion Criteria:

1. Last measurement of TSH ≥10 mU/L during levothyroxine treatment
2. Current reason for levothyroxine treatment: patients with history of thyroidectomy; radioactive iodine treatment or neck irradiation; congenital hypothyroidism; secondary hypothyroidism, or concurrent amiodarone or lithium use
3. Dose of treatment; for safety issues, patients using > 150 mcg levothyroxine per day will not be eligible
4. Concurrent treatment with liothyronine (the synthetic form of thyroid hormone T3), thiamazole, carbimazole or propylthiouracil (inhibitors of T3 and T4 synthesis).
5. Diagnosis of heart failure NYHA grade IV
6. Participation in ongoing trials of therapeutic interventions
7. Life-expectancy of less than 6 months
8. Diagnosis of dementia
9. Incapacitated adults
10. Persons that plan to move out of the region in which the study is being conducted in the next months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling participants of 60 years and older, using levothyroxine treatment, recruited from general practitioner (GP) practices in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 513 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants successfully withdrawn from levothyroxine treatment | 52 weeks after start of discontinuation
  The proportion of participants that withdraw from levothyroxine treatment successfully (defined as normal fT4 levels and TSH levels <10 mU/L) at 52 weeks after the start of the discontinuation.

SECONDARY OUTCOMES:
Proportion of participants who achieve a substantial dose reduction of levothyroxine | 52 weeks after start of discontinuation
  The proportion of participants who can achieve a substantial dose reduction of levothyroxine at 52 weeks a) defined as ≥50% and b) defined by the participants themselves
Effect of levothyroxine discontinuation on thyroid-related quality of life | 52 weeks after start of discontinuation
  Effect of levothyroxine discontinuation on thyroid-related quality of life as measured by Thyroid-specific Patient-Reported Outcome short-form (ThyPRO-39) questionnaire (range 0-100; higher scores indicate more symptoms)
Effect of levothyroxine discontinuation on general health | 52 weeks after start of discontinuation
  Effect of levothyroxine discontinuation on general health as measured by EuroQol-5D (range, -0.59 to 1.00; higher scores indicate a better quality of life)
Effect of levothyroxine discontinuation on self-rated health | 52 weeks after start of discontinuation
  Effect of levothyroxine discontinuation on general health as measured by EuroQol visual analogue scale (EQ-VAS, range 0 to 100; higher scores indicate a better quality of life)
Reflection of participants on the decision to discontinue levothyroxine treatment | 52 weeks after start of discontinuation
  Participant's view on regret after the decision to withdraw levothyroxine as measured by the Decision Regret Scale (DRS, range from 0 to 100; higher scores indicating greater regret)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobijn Gussekloo, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data can be shared upon request only, when the participant has given permission (i.e. informed consent) for data sharing concerning future research regarding thyroid disease and treatment with levothyroxine. Processed deidentified participant data such as baseline characteristics including demographic features, data on thyroid function, and data from questionnaires on secondary outcome parameters can be shared upon request. The study protocol and the statistical analysis plan (SAP) will be made available online before publication of the main results from this study. The informed consent form will be available as a supplement to the protocol paper.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: An embargo period of 2 years needs to be observed after publication of the results of the study. Thereafter, data will be available upon request for a period of 3 years.
Access Criteria: Data may be shared with researchers who provide a methodologically sound proposal. Data may be shared for individual participant data meta-analysis or for other analyses that aim to answer the research question in the approved proposal. Proposals to gain access to research data should be directed to R.K.E.Poortvliet@lumc.nl. To gain access, data requestors will need to sign a data access agreement. Data are available for 3 years at a third party website (DANS- Data Archiving and Networked Services). Authors of secondary analyses should comply with the guidelines of the International Committee of Medical Journal Editors (ICMJE).

REFERENCES:
- [Derived] Ravensberg AJ, Poortvliet RKE, Du Puy RS, Dekkers OM, Mooijaart SP, Gussekloo J. Effects of discontinuation of levothyroxine treatment in older adults: protocol for a self-controlled trial. BMJ Open. 2023 Apr 25;13(4):e070741. doi: 10.1136/bmjopen-2022-070741. PMID 37185193